CLINICAL TRIAL: NCT04196504
Title: Prevalence of Echocardioghraphic and ECG Changes in Patients With Acute Pancreatitis and Its Impact on Outcome.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaaeldin Mahmoud Ibrahim Abdelrahman, Principal Investigator, Assiut University
Other Study IDs: Echo_ECG_pancreatitis
Record Dates: First submitted 2019-10-12; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiograghy, ECG — transthoracic echocariography, 12 lead ECG

SUMMARY:
Cardiovascular system involvement with acute pancreatitis has been described before in the form of ECG changes and echocardiographic findings. However the correlation between these changes and the outcome of acute pancreatitis has not been and whether they can be used to predict mortality in these patients has been controversial.In the current study our aim is to detect echocardioghraphic and ECG changes in acute pancreatitis and investigate the significance of these changes on prognosis.

DETAILED DESCRIPTION:
Acute pancreatitis is a relatively common disease with significant morbidity and mortality. About 75% of pancreatitis is caused by gallstones or alcohol. The Atlanta classification of acute pancreatitis has been used to differentiate between severe and mild cases of acute pancreatitis. According to this classification, patients are diagnosed with severe acute pancreatitis if they show evidence of organ failure, Local complications (eg, necrosis, abscess, pseudocyst), Ranson score of 3 or higher or APACHE score of 8 or higher. Severe acute pancreatitis has a wide range of affection on nearly all body systems with various degrees of affection than affect both the clinical picture and the prognosis of the disease. the cardiovascular system involvement has been described before ,in the form of ECG changes (sinus tachycardia, arrhythmias, conduction abnormalities.. ) and echocardiographic findings (diastolic,systolic or combined dysfunction, wall motion abnormalities, pericardial effusion..). However the correlation between these changes and the outcome of acute pancreatitis has not been and whether they can be used to predict mortality in these patients has been controversial.In the current study our aim is to detect echocardioghraphic and ECG changes in acute pancreatitis and investigate the significance of these changes on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* all patients with acute pancreatitis aged more than 18 yrs admitted to Al-raghy ICU of all etiologies

Exclusion Criteria:

* patients less that 18 years
* patients above 80 years
* patients with known cardiac disease
* patients with pre-existing diabetes, chronic renal failure or malignancy.
* patients with underlying chronic pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with acute pancreatitis aged more than 18 yrs & less than 80 years old not known cardiac and with no pre-existing diabetes, chronic renal failure or malignancy with no hx of chronic pancreatitis admitted to Al-raghy ICU of all etiologies
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic (mainly diastolic dysfunction & pericardial effusion) and ECG changes (mainly QT interval) in patients with acute pancreatitis. | at admission on 1st day
  To detect the echocardiographic (mainly diastolic dysfunction & pericardial effusion) and ECG changes (mainly QT interval) in patients with acute pancreatitis.
determine the impact of these changes on outcome of patients | though out hospital admission (an average of 1 week)
  determine the impact of these changes on outcome of patients

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ashry, professor, Study Chair — Assiut University; Lobna Abdelwahid, assistant professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided